CLINICAL TRIAL: NCT00251914
Title: Supportive Test for Acid-Related Symptoms (STARS I) With Esomeprazole and a Following 7-week, Double-blind, Randomized, Placebo Controlled Treatment Period in Subjects With Upper Gastrointestinal Symptoms and With Normal Findings at Esophagogastroduodenoscopy.
Brief Title: Nexium Dyspepsia/AST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SD-NED-0021; D9610C00021
Record Dates: First submitted 2005-11-09; First posted 2005-11-11 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Gastrointestinal Disease; Signs and Symptoms, Digestive; Dyspepsia
MeSH Terms: conditions — Gastrointestinal Diseases; Signs and Symptoms, Digestive; Dyspepsia | interventions — Esomeprazole

INTERVENTIONS:
Drug: Esomeprazole

SUMMARY:
The aim is to evaluate if the resolution of upper abdominal symptoms (pain or burning) during an acid suppressive test trial of esomprazole given daily for 7 days predicts symptoms resolution at the end of a subsequent treatment period of 7 weeks.

ELIGIBILITY:
Inclusion Criteria:

* At least 3 months of symptoms of pain or burning centered in the upper abdomen prior to enrollment.
* Both Helicobacter pylori positive and negative patients eligible (Helicobacter pylori is a bacterial infection of the stomach)

Exclusion Criteria:

* Presence of clinical significant abnormal findings at the endoscopy (examination of esophagus and stomach) prior to enrollment.
* Patients with symptoms of other gastrointestinal diseases, such as Gastroesophageal Reflux Disease (GERD), Irritable Bowel Syndrome (IBS) or Inflammatory Bowel Disease (IBD).
* Helicobacter pylori eradication treatment during the last 12 months prior to enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500
Dates: Start 2002-12; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome is whether the patient is a responder or not after 8 weeks treatment.
The primary efficacy outcome is based on symptom score recorded daily during the study in a patient diary.
The patient will judge their symptoms of pain or burning centered in the upper abdomen on a four-graded scale (none, mild, moderate or severe).

SECONDARY OUTCOMES:
The secondary efficacy outcomes are whether the patient is a responder or not after 4 weeks,
The average symptom score and the percentage of symptom-free days during the 7-week treatment period,
Presence/absence of specific GI symptoms after 4 and 8 weeks of therapy

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Nexium Medical Sciences Director, MD, Study Director — AstraZeneca
Locations (215):
- Argentina (5):
  - Research Site, Buenos Aires
  - Research Site, Mendoza
  - Research Site, Rosario
  - Research Site, San Miguel de Tucumán
  - Research Site, Santa Fe
- Belgium (25):
  - Research Site, Aalst
  - Research Site, Andenne
  - Research Site, Bonheiden
  - Research Site, Bruges
  - Research Site, Brussels
  - Research Site, Brussels (Etterbeek)
  - Research Site, Brussels (Jette)
  - Research Site, Brussels (Laeken)
  - Research Site, Brussels (Woluwé-St-Lambert)
  - Research Site, Chimay
  - Research Site, Damme
  - Research Site, Edegem
  - Research Site, Eupen
  - Research Site, Genk
  - Research Site, Godinne
  - Research Site, Haine-Saint-Paul
  - Research Site, Kortenberg
  - Research Site, Kortrijk
  - Research Site, Liège
  - Research Site, Roeselare
  - Research Site, Sijsele
  - Research Site, Soignies
  - Research Site, Turnhout
  - Research Site, Wetteren
  - Research Site, Yvoir
- Brazil (9):
  - Research Site, Rio de Janeiro, Rio de Janeiro
  - Research Site, Belo Horizonte
  - Research Site, Blumenau
  - Research Site, Botucatu
  - Research Site, Campinas
  - Research Site, Florianópolis
  - Research Site, Pelotas
  - Research Site, Salvador
  - Research Site, São Paulo
- Canada (23):
  - Research Site, Edmonton, Alberta
  - Research Site, Coquitlam, British Columbia
  - Research Site, Langley, British Columbia
  - Research Site, Vancouver, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, Conception Bay South, Newfoundland and Labrador
  - Research Site, Mount Pearl, Newfoundland and Labrador
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Halifax, Nova Scotia
  - Research Site, Brampton, Ontario
  - Research Site, Courtice, Ontario
  - Research Site, Etobicoke, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, North York, Ontario
  - Research Site, Oshawa, Ontario
  - Research Site, Richmond Hill, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Windsor, Ontario
  - Research Site, Charlottetown, Prince Edward Island
  - Research Site, Montreal, Quebec
  - Research Site, Pointe-Claire, Quebec
  - Research Site, Saint-Léonard, Quebec
- Denmark (10):
  - Research Site, Aalborg
  - Research Site, Aarhus
  - Research Site, Birkerød
  - Research Site, Glostrup Municipality
  - Research Site, Hellerup
  - Research Site, Herning
  - Research Site, Holbæk
  - Research Site, København K
  - Research Site, Odense C
  - Research Site, Viborg
- France (23):
  - Research Site, Alès
  - Research Site, Angers
  - Research Site, Belfort
  - Research Site, Bois-Guillaume
  - Research Site, Cannes La Bocca
  - Research Site, Charenton-le-Pont
  - Research Site, Clermont-Ferrand
  - Research Site, Créteil
  - Research Site, Dreux
  - Research Site, Épernay
  - Research Site, Évreux
  - Research Site, Issoire
  - Research Site, Langon
  - Research Site, Lille
  - Research Site, Montélimar
  - Research Site, Nantes
  - Research Site, Narbonne
  - Research Site, Paris
  - Research Site, Rennes
  - Research Site, Saint-Denis
  - Research Site, Saint-Priest
  - Research Site, Talence
  - Research Site, Vitry-sur-Seine
- Germany (11):
  - Research Site, Cottbus, Brandenburg
  - Research Site, Saarbrücken, Saarland
  - Research Site, Dresden, Saxony
  - Research Site, Halle, Saxony-Anhalt
  - Research Site, Magdeburg, Saxony-Anhalt
  - Research Site, Berlin
  - Research Site, Biederitz
  - Research Site, Leipzig
  - Research Site, Magdeburg
  - Research Site, Mandelbachtal-Ommersheim
  - Research Site, Potsdam
- Greece (3):
  - Research Site, Athens
  - Research Site, Piraeus
  - Research Site, Thessaloniki
- Iceland (2):
  - Research Site, Hafnarfjördur
  - Research Site, Reykjavik
- Italy (20):
  - Research Site, San Benedetto del Tronto, AP
  - Research Site, L’Aquila, AQ
  - Research Site, Biella, BI
  - Research Site, Brescia, BS
  - Research Site, San Cataldo, CL
  - Research Site, Como, CO
  - Research Site, Cremona, CR
  - Research Site, Catania, CT
  - Research Site, Milan, MI
  - Research Site, Pisa, PI
  - Research Site, Reggio Calabria, RC
  - Research Site, Roma, Roma
  - Research Site, Sondalo, SO
  - Research Site, Sondrio, SO
  - Research Site, Torino, TO
  - Research Site, San Daniele del Friuli, UD
  - Research Site, Udine, UD
  - Research Site, Bologna
  - Research Site, Castellammare di Stabia
  - Research Site, Torre del Greco
- Norway (37):
  - Research Site, Aksdal
  - Research Site, Arendal
  - Research Site, Bergen
  - Research Site, Brumunddal
  - Research Site, Bøverbru
  - Research Site, Eidehavn
  - Research Site, Elverum
  - Research Site, Fevik
  - Research Site, Fitjar
  - Research Site, Flatåsen
  - Research Site, Fredrikstad
  - Research Site, Fyllingsdalen
  - Research Site, Hafrsfjord
  - Research Site, Hafslundsøy
  - Research Site, Hamar
  - Research Site, Heimdal
  - Research Site, Høvik
  - Research Site, Jessheim
  - Research Site, Kokstad
  - Research Site, Kolbjørnsvik
  - Research Site, Langesund
  - Research Site, Larvik
  - Research Site, Løten
  - Research Site, Løvenstad
  - Research Site, Moss
  - Research Site, Nesttun
  - Research Site, Oslo
  - Research Site, Paradis
  - Research Site, Rasta
  - Research Site, Rolvsøy
  - Research Site, Ski
  - Research Site, Sogndal
  - Research Site, Spydeberg
  - Research Site, Stjørdal
  - Research Site, Svelvik
  - Research Site, Sørumsand
  - Research Site, Trondheim
- Romania (4):
  - Research Site, Brasov
  - Research Site, Bucharest
  - Research Site, Târgu Mureş
  - Research Site, Tg. Mures
- Research Site, Singapore, Singapore
- South Africa (8):
  - Research Site, Bloemfontein
  - Research Site, Cape Town
  - Research Site, Durban
  - Research Site, Johannesburg
  - Research Site, Lyttelton Manor
  - Research Site, Parktown
  - Research Site, Pretoria
  - Research Site, Tygerberg
- Spain (6):
  - Research Site, Santiago, A Coruña
  - Research Site, Santiago de Compostela, A Coruña
  - Research Site, Barcelona, Barcelona
  - Research Site, Viladecans, Barcelona
  - Research Site, Madrid, Madrid
  - Research Site, Seville, Sevilla
- Sweden (21):
  - Research Site, Arbrå
  - Research Site, Ängelholm
  - Research Site, Gothenburg
  - Research Site, Gullspång
  - Research Site, Höganäs
  - Research Site, Jönköping
  - Research Site, Kristinehamn
  - Research Site, Lund
  - Research Site, Malmo
  - Research Site, Rättvik
  - Research Site, Skövde
  - Research Site, Södertälje
  - Research Site, Stockholm
  - Research Site, Sundsbruk
  - Research Site, Täby
  - Research Site, Trollhättan
  - Research Site, Uddevalla
  - Research Site, Upplands Vasby
  - Research Site, Varberg
  - Research Site, Värnamo
  - Research Site, Västerås
- Switzerland (7):
  - Research Site, Baden, Canton of Aargau
  - Research Site, Frick, Canton of Aargau
  - Research Site, Spreitenbach, Canton of Zurich
  - Research Site, Basel
  - Research Site, Ennetbaden
  - Research Site, Sankt Gallen
  - Research Site, Sargans

REFERENCES:
- [Derived] Paggi S, Radaelli F, Amato A, Meucci G, Mandelli G, Imperiali G, Spinzi G, Terreni N, Lenoci N, Terruzzi V. The impact of narrow band imaging in screening colonoscopy: a randomized controlled trial. Clin Gastroenterol Hepatol. 2009 Oct;7(10):1049-54. doi: 10.1016/j.cgh.2009.06.028. Epub 2009 Jul 1. PMID 19577008
- [Derived] Talley NJ, Vakil N, Lauritsen K, van Zanten SV, Flook N, Bolling-Sternevald E, Persson T, Bjorck E, Lind T; STARS I Study Group. Randomized-controlled trial of esomeprazole in functional dyspepsia patients with epigastric pain or burning: does a 1-week trial of acid suppression predict symptom response? Aliment Pharmacol Ther. 2007 Sep 1;26(5):673-82. doi: 10.1111/j.1365-2036.2007.03410.x. PMID 17697201